CLINICAL TRIAL: NCT00676793
Title: Phase II Clinical Trial to Determine if Polyphenon E Inhibits c-Met Signaling and Activation of Pathways Contributing to Breast Cancer Progression
Brief Title: A Study of the Effect of Polyphenon E (Green Tea Extract) on Breast Cancer Progression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Jerry McLarty, Professor, Louisiana State University Health Sciences Center Shreveport
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H04-179
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; EGCG; Polyphenon E; c-Met; VEGF; HGF
MeSH Terms: conditions — Breast Neoplasms | interventions — polyphenon E

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Polyphenon E (Experimental): This is a single arm study comparing changes within patients before and after receiving the experimental drug Polyphenon E for the duration of the study, between recruitment and surgery for breast cancer.
  Interventions: Drug: Polyphenon E

INTERVENTIONS:
Drug: Polyphenon E — Four 200mg capsules daily taken with a meal, for the duration of the study.

SUMMARY:
To see if an extract of green tea can affect certain markers of breast cancer and breast cancer progression in women with a recent biopsy positive for cancer and who are scheduled for surgery.

DETAILED DESCRIPTION:
To evaluate the short-term effects of a daily dose of Polyphenon E administered during the interval between breast biopsy and surgery in women with recently diagnosed breast cancer. Endpoints will be changes in serum and tissue biomarkers related to progression of cancer.

The effect of Polyphenon E on tumor cell c-Met expression and phosphorylation is the primary objective. Secondary objectives include the effects on the other tissue and serum biomarkers. Evaluation of the safety and tolerability of Polyphenon E in this subject population is another objective.

1.1 Determine the effects of Polyphenon E on tumor cell c-Met expression and phosphorylation levels in patients with breast cancer

1.2 Determine the effects of Polyphenon E on PI-3K activation in patients with breast cancer

1.3 Determine the effects of Polyphenon E on MAPK activation in patients with breast cancer

1.4 Determine the effects of Polyphenon E on expression levels of other proteins involved in motility and invasion such as Rho GTPases and extracellular proteinases in patients with breast cancer

1.5 Determine the effects of Polyphenon E on markers of angiogenesis in patients with breast cancer

1.6 Determine the effects of Polyphenon E on other serum markers: C-reactive protein (CRP), Insulin-Like Growth factor I (IGF-I), Insulin-like Growth Factor Binding Protein 3 (IGFBP-3) and Hepatocyte Growth Factor HGF

1.7 Evaluate the safety and tolerability of Polyphenon E in this subject population

ELIGIBILITY:
Inclusion Criteria:

* Definitive biopsy demonstrating primary breast cancer
* Residual breast cancer requiring additional surgical resection
* Stage I, II or III disease
* Patient has ability to give signed informed consent
* Normal hepatic and renal function (creatinine<1.5, transaminases <1.5 times upper limit of normal).
* ECOG Performance status of 0 or 1.
* Age ≥ 21 years and less than 75

Exclusion Criteria:

* Prior hormonal or surgical therapy for breast cancer
* Abnormal liver function test
* Liver or kidney problems that would interfere with metabolism of study drug
* Any condition that would hamper informed consent or ability to comply with study protocol
* Participation in another research study in the last three months
* Known malignancy at any site other than breast
* Recent consumption of green tea (5 or more cups per day, within one week prior to biopsy)
* Allergy or intolerance to any component of green tea
* Inability or refusal to comply with definitive surgical therapy

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-05; Primary Completion 2009-12 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Burton, M.D., Principal Investigator — LSU Health Sciences Center Shreveport
Locations (2):
- United States (2):
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Columbia Presbyterian Hospital, New York, New York

REFERENCES:
- [Result] Proffered Oral Presentations - Intervention Studies Abstract PR-05: Effects of presurgical administration of tea polyphenols in women with operable breast cancer Julie L. Campbell1, James Cardelli2, Jerry McLarty2, Dawn Hershman1, Bret Taback1, Susan Refice1, Stephanie Wang2, Rebecca Bigelow2 and Katherine Crew1 1Columbia University Medical Center, New York, NY 2Louisiana State University Health Sciences Center, Shreveport, LA Cancer Prevention Research: December 2010; Volume 3, Issue 12, Supplement 2. doi: 10.1158/1940-6207.PREV-10-PR-05

RESULTS

PARTICIPANT FLOW:
Groups:
- ECGC and Breast Cancer: Single arm for a phase II study of EGCG extract and breast cancer. Subjects are asked to take 4 polyphenol E (200mg) capsules daily with a meal for the duration of the study. Biomarkers are measured at baseline and then again at presurgery, the end point for the study.
Period: Overall Study
Arm/Group | ECGC and Breast Cancer
Started | 32
Completed | 19
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | ECGC and Breast Cancer
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum VEGF in Breast Cancer
Description: Change in serum VEGF from baseline to post treatment with polyphenon E.
Time Frame: Baseline and 4 to 6 weeks
Population: Number of participants for analysis was determined per protocol.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | ECGC and Breast Cancer
Number analyzed (Participants) | 19
pg/ml | 270 [-142.5 to 581.25]
Statistical Analysis 1: Comparison: ECGC and Breast Cancer; The null hypothesis is that there is no change, i.e. median change=0.0; Test type: Superiority or Other; p = 0.078, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Serum HGF and Breast Cancer
Description: Change in serum HGF from baseline to post Polyphenol E treatment.
Time Frame: Baseline and 4 to 6 weeks
Population: Number of participants for analysis was determined per protocol.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- ECGC and Breast Cancer: The effect of ECGC extract on biomarkers in breast cancer.
Arm/Group | ECGC and Breast Cancer
Number analyzed (Participants) | 19
pg/ml | 155.0 [-143.75 to 700.625]
Statistical Analysis 1: Comparison: ECGC and Breast Cancer; The null hypothesis is that there is no change, i.e. median change=0.0; Test type: Superiority or Other; p = 0.094, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | ECGC and Breast Cancer
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 3/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECGC and Breast Cancer (N=32)
Stomach Cramps (Gastrointestinal disorders) | 2 (2)
Increase in amylase and lypase (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No